CLINICAL TRIAL: NCT05977205
Title: The Impact of Self-quarantining on Glycemic Control, Diabetes Self-management and Distress During the Coronavirus Outbreak
Brief Title: COVID-19 Glycemic Control Study
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Eelco JP de Koning, Principal Investigator, Professor in Diabetology, Leiden University Medical Center
Other Study IDs: NL73778.058.20
Record Dates: First submitted 2023-07-31; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: COVID-19 Pandemic; Type 1 Diabetes; Type 2 Diabetes; Beta Cell Transplantation; Social isolation; Glycemic control; Distress; COVID-19 Lockdown
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; COVID-19; Social Isolation | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 1 Diabetes: 280 patients with type 1 diabetes
  Interventions: Other: No interventions, observational study
- Type 2 Diabetes: 155 patients with type 2 diabetes
  Interventions: Other: No interventions, observational study
- Type 1 Diabetes with Islet or Pancreas Transplantation: 23 patients with islet transplantation, 7 with pancreas transplantation, 27 with simultaneous pancreas-kidney transplantation
  Interventions: Other: No interventions, observational study

INTERVENTIONS:
Other: No interventions, observational study — Not applicable, no interventions, observational study

SUMMARY:
Diabetes mellitus is a chronic disease characterized by the inability of the body to maintain normoglycemia. Treatment of diabetes relies mostly on diabetes self-management, requiring a large investment of time and energy on a daily basis. Psychological wellbeing, behavioral patterns and social context play a major role in diabetes self-management and glycemic control. Social isolation behavior (self-quarantining) may impact glycemic control by influencing daily routines, therapy adherence, physical activity, and self-measurement and eating behaviors. Therefore, a period of nationwide self-quarantine, such as during the lockdown issued during the COVID-19 outbreak in the Netherlands, may have a large effect on glycemic control in patients with diabetes.

In this observational cross sectional study, we aim to assess the impact of long-term self-quarantine on glycemic control, diabetes self-management and distress in patients with type 1 and type 2 diabetes mellitus.

A specific subgroup of patients with T1D are those with complicated diabetes who have received a pancreas or islet transplantation and use immunosuppression, having multiple risk factors for severe COVID-19. The impact of lockdown strategies on mental and physical health is expectedly even greater in patients at even higher risk for severe COVID-19. We therefore additionally investigated differences in behavioral, mental and physical implications of a nationwide lockdown on patients with type 1 diabetes with and without islet or pancreas transplantation.

Measurements will be performed during the lockdown period. Patients will be asked to perform a fingerprick HbA1c measurement once, sent back to the LUMC by mail. Data from continuous or flash glucose monitoring devices will be collected according to standard clinical practice. Furthermore, patients will be asked to fill out an online questionnaire once on diabetes self-management behavior, well-being and distress, along with questions about health status, level of education, medication use, employment, social situation and the impact of self-quarantine on daily routines. In this questionnaire, we ask patients to compare certain aspects of their life (e.g. anxiety, stress, weight, physical activity, glycemic control) at the time of the lockdown to before the lockdown. Data on demographics, type of diabetes, weight, BMI and HbA1c prior to the COVID-19 outbreak will be derived from the patient's electronic health file.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with type 1 or type 2 diabetes
* Ability to perform fingerpricks
* Sufficient comprehension of the Dutch language
* Ability to fill out online questionnaires

Exclusion Criteria:

* Pregnancy
* Newly diagnosed malignancy, with the exclusion of non-melanoma skin cancer, in the previous 6 months
* Chemotherapy or immunotherapy for malignancy
* Admission to hospital or rehabilitation center

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes (with and without islet or pancreas transplantation) and type 2 diabetes, recruited from the diabetes outpatient clinic of the LUMC.
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Glycemic control | HbA1c measurement during lockdown (8 - 11 weeks after the start of the lockdown (March 15th 2020)) compared to last measurement before lockdown (last known measurement before March 15th 2020)
  HbA1c (mmol/mol Hb)

SECONDARY OUTCOMES:
Glycemic control | 2 week period during lockdown compared to 2 week period before lockdown
  Continuous Glucose Measurement parameters (time in range, time above range, time below range)
Stress | PSS During lockdown + self-comparison change to before lockdown (questionnaire filled in between 8 - 11 weeks after the start of the lockdown (March 15th 2020))
  Perceived Stress Scale (PSS) + self-reported change in stress during lockdown compared to before lockdown
Anxiety | Questionnaire filled in between 8 - 11 weeks after the start of the lockdown (March 15th 2020))
  Self-reported change in anxiety during lockdown compared to before lockdown
Weight | Questionnaire filled in between 8 - 11 weeks after the start of the lockdown (March 15th 2020))
  Self-reported weight change during lockdown compared to before lockdown
Physical activity | Questionnaire filled in between 8 - 11 weeks after the start of the lockdown (March 15th 2020))
  Self-reported change in physical activity during lockdown compared to before lockdown
Glycemic control and insulin requirements | Questionnaire filled in between 8 - 11 weeks after the start of the lockdown (March 15th 2020))
  Self-reported change in difficulty with glycemic control and insulin requirements during lockdown compared to before lockdown
Social isolation behaviour | Questionnaire filled in between 8 - 11 weeks after the start of the lockdown (March 15th 2020))
  Self-reported social isolation behaviour during lockdown
Fear of COVID-19 infection | Questionnaire filled in between 8 - 11 weeks after the start of the lockdown (March 15th 2020))
  Fear of contracting COVID-19, scored using a Visual Analogue Scale (1-10), during lockdown

CONTACTS AND LOCATIONS:
Overall Officials: Eelco JP de Koning, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Landstra CP, Ruissen MM, Regeer H, Nijhoff MF, Ballieux BEPB, van der Boog PJM, de Vries APJ, Huisman SD, de Koning EJP. Impact of a Public Health Emergency on Behavior, Stress, Anxiety and Glycemic Control in Patients With Pancreas or Islet Transplantation for Type 1 Diabetes. Transpl Int. 2024 Mar 27;37:12278. doi: 10.3389/ti.2024.12278. eCollection 2024. PMID 38601276

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT05977205/Prot_ICF_000.pdf